CLINICAL TRIAL: NCT00162838
Title: Effects of Periodontal Pathogens, Porphyromonas Gingivalis and Tannerella Forsythensis, on Cytokine Production From Human Monocyte-Derived Dendritic Cells.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9261700824; NTUH-93S039
Record Dates: First submitted 2005-09-12; First posted 2005-09-13 (Estimated); Last update posted 2005-11-23 (Estimated); Status verified 2003-05

CONDITIONS: Periodontal Disease
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Periodontitis develops due to subgingival infection with specific microbial pathogen from dental plaque. The bacteria can activate immunoinflammatory mechanisms within the local periodontal tissues that lead to destruction of collagen and alveolar bone. Human gingiva contains Langerhans and connective tissue dendritic cells. Signals from periodontal pathogen can induce dendritic cells to maturation,rapidly increasing surface expression of MHC class II, costimulatory molecules, and secrete proinflammatory cytokines to regulate adaptive T cell immune response. Studies on cytokines have led to controversy about different T cell subsets associated with the progression of periodontitis. Seymour proposed that susceptibility to periodontal disease progression involve a predominantly Th2 response while Ebersole speculated that Th2 cells providing protective function. It is possible that a given pathogen may produce different maturation signals by activating DCs induce a given type of immune response. In this study, we observed the profiles and amounts of cytokine production of DCs stimulated with P. gingivalis and T. forsythensis compared with E. coli, to see whether the periodontal pathogens may induce different response of dendritic cells in the innate immunity.

DETAILED DESCRIPTION:
Periodontitis develops due to subgingival infection with specific microbial pathogen from dental plaque. The bacteria can activate immunoinflammatory mechanisms within the local periodontal tissues that lead to destruction of collagen and alveolar bone. Bacterial antigens can release from the supra and subgingival dental plaque on the tooth surface as well as from bacteria attached to mucosal surfaces. The sulcular epithelium served as a physical barrier to the insult of the bacteria, the presence of Langerhans cells is also responsible for communication with the immune system. Dendritic cells (DCs), the most effective antigen-presenting cells, contact and process the antigens. Signals from pathogen induce dendritic cells to maturation. Mature DCs rapidly increase surface expression and stability of MHC class I and class II-peptide complexes, upregulate the surface expression of adhesion and co-stimulatory molecules (CD40, CD54, CD80, and CD86) and secrete proinflammatory cytokines such as IL-1, IL-6, IL-12…….. then they migrate to lymphoid organs, where they regulate T cell immune response. Human gingiva contains Langerhans and connective tissue dendritic cells. Immature dendritic cells appeared to be limited to the epithelium, whereas mature dendritic cells were restricted to the connective tissue. Studies on cytokines have led to controversy about the the different T cell subsets associated with the progression of periodontitis. Seymour proposed that susceptibility to periodontal disease progression involve a predominantly Th2 response while Ebersole speculated that Th2 cells providing protective function. Progression of periodontitis is also associated with the presence of gram-negative anaerobic microorganism such as Porphyromonas gingivalis, Bacteroides forsythus. Different bacteria and their LPS can elicit strikingly different response. It is possible that a given pathogen may produce different maturation signals by selectively activating a particular DC subset to induce a given type of immune response. In this study, we observed the profiles and amounts of cytokine production of DCs stimulated with P. gingivalis and T. forsythensis compared with E. coli, to see whether the periodontal pathogens may induce different response of dendritic cells in the innate immunity.

ELIGIBILITY:
Inclusion Criteria:

* Healthy

Exclusion Criteria:

-

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2003-10

CONTACTS AND LOCATIONS:
Overall Officials: Man-ying Wong, DDS, MS, Principal Investigator — Department of Periodontics, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan